CLINICAL TRIAL: NCT01380808
Title: A Phase II Study of Capecitabine and Pseudomonas Aeruginosa Combination in the Salvage Treatment of Metastatic Breast Cancer
Brief Title: Capecitabine and Pseudomonas Aeruginosa Combination in Metastatic Breast Cancer (MBC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xichun Hu, Dr, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Fudan BR2011-05
Record Dates: First submitted 2011-05-10; First posted 2011-06-27 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2013-07

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- experimental arm (Experimental): capecitabine and pseudomonas aeruginosa combination
  Interventions: Drug: capecitabine and pseudomonas aeruginosa combination

INTERVENTIONS:
Drug: capecitabine and pseudomonas aeruginosa combination — capecitabine 1000mg/m2 bid, po. pseudomonas aeruginosa 0.5ml loading dose,1ml qod ih.
  Other Names: capecitabine; pseudonomas aeruginosa

SUMMARY:
The progression free survival could be prolonged adding pseudomonas aeruginosa to monotherapy capecitabine.

DETAILED DESCRIPTION:
the efficacy of the combination is much better than monotherapy

ELIGIBILITY:
Inclusion Criteria:

1. Female between 18 and 70 years old
2. Patients with histologic proved metastatic breast cancer, unsuitable to be treated locally.
3. Patients with Her-2 negative breast cancer(HER-2 negative or one plus by IHC test , if HER-2 two plus by IHC,FISH result should be negative)
4. Disease progression after anthracycline and/or taxane regimen therapy and candidate for capecitabine monotherapy
5. Patients previously treated by capecitabine containing regimen should response to the chemotherapy containing capecitabine and progressed at least 4 months after the last capecitabine treatment
6. Karnofsky score more than 70；ECOG 0~2；
7. Normal functions with heart, liver,renal and bone marrow
8. WBC≥4×109/L；Hb≥90 g/L；plt≥100×109/L
9. Got ICF before enrollment

Exclusion Criteria:

1. Pregnant or breast-feeding women or positive serum pregnancy test
2. Uncontrolled brain metastases. Patients with brain metastases must be locally treated and the disease must be stable for at least one month at the time of enrolling
3. Participation in any investigational drug study within 4 weeks preceding treatment start.
4. Concurrent other malignancy at other sites or previous other cancer within the last 5 years, with the exception of adequately treated in situ carcinoma of cervix uteri or basal or squamous cell carcinoma of the skin or a contralateral breast cancer.
5. Serious uncontrolled intercurrent infections
6. Poor compliance

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
progression free survival | 1 year

SECONDARY OUTCOMES:
overall response rate | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, MD,PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, China

REFERENCES:
- [Derived] Lv F, Cao J, Liu Z, Wang Z, Zhang J, Zhang S, Wang L, Zhao X, Shao Z, Wang B, Hu X. Phase II study of Pseudomonas aeruginosa-Mannose-Sensitive hemagglutinin in combination with capecitabine for Her-2-negative metastatic breast cancer pretreated with anthracycline and taxane. PLoS One. 2015 Mar 13;10(3):e0118607. doi: 10.1371/journal.pone.0118607. eCollection 2015. PMID 25768439